CLINICAL TRIAL: NCT06859502
Title: "Registro Dati Nazionale Dell'Istituto Virtuale Delle Malattie Cerebrovascolari" "National Database of the Virtual Institute of Cerebrovascular Diseases"
Brief Title: National Database of the Virtual Institute of Cerebrovascular Diseases
Acronym: BIG-MENTI
Status: Recruiting | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: BIG-MENTI
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-04

CONDITIONS: Cerebrovascular Disease
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with cerebrovascular diseases: Participants will be recruited at any stage of cerebrovascular disease management: acute hospitalization, subsequent neuromotor rehabilitation, or follow-up outpatient visit three months after the acute event.

SUMMARY:
The overall objective of the study is to identify prognostic predictors of cerebrovascular disease during various stages of the cerebrovascular disease itself, namely: hospitalization at the acute care facility, residential hospitalization at neurorehabilitation facilities, outpatient follow-up visits, and day hospital admissions at the various facilities. The aim is to obtain data on those factors that can influence the prognosis, thus the clinical outcome, of patients with cerebrovascular disease.

Cerebrovascular diseases are defined by the World Health Organization (WHO) as "all those disorders in which there is an area of the brain transiently or permanently affected by ischemia or bleeding or in which one or more cerebral blood vessels are primarily affected in a pathological process, or a combination of the two conditions mentioned above." These diseases include a wide range of conditions, of which ischemic stroke and cerebral hemorrhage are the most common. Given the high overall frequency of these diseases and, consequently, the high social and economic cost of them on the population, it is essential to recognize as soon as possible those factors capable of predicting the time course of patients affected, as you are, by these diseases, also with a view to identifying strategies to improve the prognosis of patients for whom an unfavorable outcome is predicted. In addition, given the high prevalence of cerebrovascular disease, it is necessary that an extremely large patient population be enrolled, and thus an enormous amount of data be collected, in order for meaningful results to be obtained.

The primary objective of this study is, in fact, to collect a large amount of clinical data, i.e., to establish a national data registry, obtained from the records of patients with cerebrovascular diseases that began after January 1, 2016, in order to be able to identify and define the subtypes of each cerebrovascular disease associated with poor prognosis. The secondary objectives are to identify clinical, neurophysiological, radiological, and biomarker data that are able to predict the clinical course of cerebrovascular disease over time and to identify prognostic scores obtained from the combination of the variables first indicated. With this study, we also aim to identify those clinical, radiological, and neurophysiological data that are able to help the clinician in the early differential diagnosis of these diseases and that are able to predict the occurrence of spontaneous or procedure-related complications and the successful outcome of treatment. Finally, we aim to identify those clinical, radiological, and neurophysiological variables that are able to predict a good outcome of rehabilitation performed as a result of the onset of cerebrovascular disease.

DETAILED DESCRIPTION:
Considering the high incidence of cerebrovascular diseases, it therefore seems obvious how, in order to be able to demonstrate causal links and to search for prognostic factors with a high level of evidence, a systematic collection of large-scale data involving different facilities scattered throughout the country is necessary. Such systematic collection would allow both, as just mentioned, to obtain valid data on high-prevalence diseases, such as stroke, and to obtain sufficient evidence for the diagnostic and prognostic framing of those cerebrovascular diseases with lower incidence. In addition, considering the large amount of data, it seems clear that there is a need for a rapid and efficient information collection system that can guarantee an optimal result without overburdening the work of healthcare personnel. In this context, in 2017 the Ministry of Health established the IRCCS Network of Neuroscience and Neurorehabilitation (RIN).

Within this framework, numerous Virtual Institutes, specialized by disease areas, are being developed in a cross-cutting manner to provide the Network with its own strong identity, harmonize IRCCS activities, rationalize investments and resources, build large cohorts, and interact with international networks. To this end, a survey was sent to all Network members in October 2020 to indicate, in the specific area of Cerebrovascular Diseases: the human, infrastructural and technological resources available; and the volume and type of specific clinical activity carried out in the year 2019.

Thirty-two centers responded to the survey, expressing interest in the participation of the forming Virtual National Institute (IVN) of Cerebrovascular Diseases. The geographical distribution of participating centers is as follows: 22 in the North, 6 in the Center and 4 in the South. Peculiarities of this IVN are the high volume of patients with such frequent diseases, the great clinical specialization, the high technological level of care at all stages of the disease, and the required and necessary dynamism and timeliness of intervention.

The individual members of this IVN possess a great and diverse expertise in both care activities and clinical and pre-clinical research. In addition, considering the high sociomedical burden of the set of these pathologies, largely related to the permanent disability they entail, the IVN of Cerebrovascular Diseases will have the peculiarity of being able to follow the entire pathway of the Patient from the acute phases (hospital) to those of rehabilitation (in neurorehabilitation centers) until the return home. Through this study, the aim is to create a national registry for these diseases.

The primary objective of the study is to identify and define the various subtypes of each cerebrovascular disease falling under the following codes of the International Classification of Diseases, 9th revision (ICD-9): ICD-9 430-438, associated with poor prognosis.

Secondary objectives:

* Identification of clinical variables of each cerebrovascular pathology correlated with the prognosis of the same;
* Identification of biomarkers of each cerebrovascular pathology correlated with the prognosis of the same;
* Identification of the radiological variables of each cerebrovascular pathology correlated with the prognosis of the same;
* Identification of neurophysiological variables of each cerebrovascular pathology correlated with the prognosis of the same;
* Identification of prognostic scores for each cerebrovascular disease based on the combination of clinical, radiological, neurophysiological and biomarker variables;
* Identification of the clinical, radiological and neurophysiological variables and biomarkers of each cerebrovascular disease that will help the clinician in early differential diagnosis;
* Identifications of the clinical, radiological, and neurophysiological variables and biomarkers of each cerebrovascular pathology that can predict the development of spontaneous or procedure-related complications of treatment;
* Identifications of the clinical, radiological, and neurophysiological variables and biomarkers of each cerebrovascular pathology capable of predicting the successful outcome of pharmacological or procedural therapies;
* Identification of clinical, radiological, and neurophysiological variables and biomarkers of each cerebrovascular pathology useful for personalization of rehabilitation treatment and able to predict good functional outcome following the same rehabilitation treatments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebrovascular pathology defined according to the 1990 NINDS special report2 as "all disorders in which an area of the brain is transiently or permanently affected by ischemia or bleeding and/or in which one or more of the blood vessels of the brain are primarily altered by a pathological process," falling under the following International Classification of Diseases, 9th revision (ICD-9) codes: ICD-9 430-438;
* Informed consent provided by the patient or the patient's legal representative in the case of incapacitation, or by the parents/guardians in the case of minor subjects.

Exclusion Criteria:

* The patient, his or her legal representative in the case of incapacitation, or his or her parents/guardians in the case of minor subjects irrefutably express the will to leave the study;
* Onset of cerebrovascular disease before January 1, 2016.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited at each individual center by the principal investigator (PI) or one of the local sub-investigators (sub-I) at any stage of cerebrovascular disease management: acute hospitalization, subsequent neuromotor rehabilitation, or follow-up outpatient visit three months after the acute event.
Sampling Method: Non-Probability Sample
Enrollment: 312800 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2053-04-01 (Estimated); Study Completion 2054-04-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | From enrollment to maximum 1 month
  Identification and definition of the various subtypes of each cerebrovascular disease, falling under the following International Classification of Diseases, 9th revision (ICD-9) codes: ICD-9 430-438, associated with poor prognosis.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Don Gnocchi, Florence, FI, Italy

IPD SHARING:
Plan to Share IPD: Undecided